CLINICAL TRIAL: NCT02321215
Title: Effectiveness and Feasibility of Delivering an Introductory Education Program to Patients Admitted to Hospital With an Acute Exacerbation of COPD - a Pilot Randomized Controlled Trial
Brief Title: Effectiveness and Feasibility of Delivering an Education Program to Patients With an Acute Exacerbation of COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Tania Janaudis Ferreira, Scientist, West Park Healthcare Centre
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CRHP_EducationAECOPD2014
Record Dates: First submitted 2014-12-03; First posted 2014-12-22 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Obstructive Pulmonary Disease With (Acute) Exacerbation
Keywords: AECOPD; COPD; education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Usual care: This group will receive usual care from their physician without any special focus on education. At the end of the study period, patients that were assigned to the control group will receive the booklet at home and be offered two education sessions by phone or in-person if the patient is willing to return to the hospital.
- Education Intervention (Active Comparator): Introductory disease education: This group will attend two one-on-one education sessions. The educational content will be standardized and a checklist will be used to ensure that all topics are addressed. The sessions will focus on enhancing self-efficacy in areas that are thought to be important to individuals who recently had an AECOPD.
  Interventions: Other: Introductory Disease Education

INTERVENTIONS:
Other: Introductory Disease Education — This intervention will consist of two one-on-one education sessions, each lasting 30 minutes.
  Other Names: COPD Education Program
  Arms: Education Intervention

SUMMARY:
The purpose of this study is to determine if it is effective and feasible to provide a chronic obstructive pulmonary disease (COPD) education program to patients admitted with an acute exacerbation of COPD.

DETAILED DESCRIPTION:
Following an acute exacerbation of chronic obstructive pulmonary disease (AECOPD) evidence strongly suggests that all patients should be discharged with an action plan, consisting of identified patient responsibilities for their ongoing care and advice on recognizing and seeking help in the event of future acute exacerbations. Despite these recommendations, structured chronic obstructive pulmonary disease (COPD) specific education is rarely offered within acute hospital settings and, in addition, research in this area is limited. This study aims to determine the effectiveness and feasibility of an introductory education program delivered during and shortly after an AECOPD hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* medically confirmed diagnosis of AECOPD (alone or combined with other conditions)
* capable of understanding the study information and giving informed consent

Exclusion Criteria:

* admitted due to lung diseases other than COPD
* received COPD education in the previous 6 months (in primary care, acute or rehabilitation hospitals)
* presence of diagnosis of dementia or incapacity to learn due to cognitive issues
* have medical, cognitive or language limitations to communicating in written or spoken English
* have participated or been asked to participate in the trial before
* in the intensive care unit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in disease specific knowledge | This primary outcome measure will be collected prior to randomization and approximately four weeks after admission
  Bristol COPD Knowledge Questionnaire (BCKQ)
Change from baseline in information needs | This primary outcome measure will be collected prior to randomization and approximately four weeks after admission
  Lung Information Needs Questionnaire (LINQ)

SECONDARY OUTCOMES:
Feasibility measure: number of eligible patients | This outcome variable will be noted within 1-2 days of hospital admission with an AECOPD (when determining patient eligibility, before randomization).
Feasibility measure: ease of recruiting patients | This outcome variable will be noted within 1-2 days of hospitalization, while the patient is being recruited (before randomization).
  Questions: (1) Is it easy to locate the patient in their room? (Yes/No) (2) How many times did the RA try to find the patient in the room before successfully finding them there? (#) (3) Does the patient have enough time to meet with the RA? (Yes/No)
Feasibility measure: compliance to the sessions | This outcome measure will be noted after each education session. The education sessions will take place between 3-15 days after hospital admission for an AECOPD. Two education sessions will be delivered to every patient enrolled in the intervention arm.
  Questions: (1) Is the participant able to complete the half-hour session? (Yes/No) (2) How many times was the education session interrupted for any reason? (#)
Feasibility measure: follow-up rates | This outcome variable will be noted between days 20-30 following admission to hospital (approximately four weeks after hospital admission).
  Proportion of subjects that complete the follow up stage (questionnaire responses)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Goldstein, MD, Study Chair — West Park Healthcare Centre; Samantha Harrison, PhD, Study Chair — West Park Healthcare Centre; David Fishbein, MD, Study Chair — Humber River Hospital; Sean Carr, MD, Study Chair — Humber River Hospital; Andrea Gershon, MD, Study Chair — Sunnybrook Health Sciences Centre
Locations (1):
- Humber River Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Janaudis-Ferreira T, Carr SJ, Harrison SL, Gershon AS, Milner SC, Carr S, Fishbein D, Goldstein R. Can Patients With COPD Assimilate Disease-Specific Information During an Acute Exacerbation?: Results of a Pilot Randomized Controlled Trial. Chest. 2018 Sep;154(3):588-596. doi: 10.1016/j.chest.2018.05.028. Epub 2018 Jun 4. PMID 29879395